CLINICAL TRIAL: NCT01349751
Title: Clinical Characteristics of Spinal Levobupivacaine: Hyperbaric Compared With Isobaric Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Vimolluck Sanansilp, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: SiEC 197/2549
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Observation of Neuromuscular Block; Disease (or Disorder); Gynecological
Keywords: abdominal incision; hyperbaric; isobaric; levobupivacaine; spinal anaesthesia
MeSH Terms: conditions — Disease | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- isobaric levobupivacaine (Active Comparator): spinal isobaric levobupivacaine
  Interventions: Drug: isobaric levobupivacaine
- hyperbaric levobupivacaine (Active Comparator): hyperbaric levobupivacaine
  Interventions: Drug: hyperbaric levobupivacaine

INTERVENTIONS:
Drug: isobaric levobupivacaine — 0.42% either isobaric levobupivacaine 3 ml spinal injection once
  Other Names: Chirocaine, Abbott Laboratories, Nycomed Pharma AS, Norway
  Arms: isobaric levobupivacaine
Drug: hyperbaric levobupivacaine — 0.42% hyperbaric levobupivacaine 3 ml spinal injection once
  Other Names: Chirocaine, Abbott Laboratories, Nycomed Pharma AS, Norway
  Arms: hyperbaric levobupivacaine

SUMMARY:
The authors would like to investigate the blocking characteristics, surgical quality and side effects of intrathecal levobupivacaine whether there are any differences between the hyperbaric and the isobaric formulation for gynaecologic surgeries which need higher block level than the urological surgeries.

DETAILED DESCRIPTION:
The investigators study in the similar patients, give the same intervention except the baricity of levobupivacaine. The investigators record the level of sensory block and modified Bromage score for motor blockade.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III, aged 18-70 yr, scheduled for elective gynaecologic surgery, (total abdominal hysterectomy (TAH), TAH with uni-/bilateral salpingo-oophorectomy (SO), uni-/bilateral ovarian cystectomy, or myomectomy

Exclusion Criteria:

* contraindications for spinal block, body mass index (BMI) more than 35 kg/m2 and height less than 150 cm

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
time to T4-dermatome sensory blockade | 30 minutes
  to investigate specific blocking characteristics of intrathecal hyperbaric levobupivacaine compared with isobaric levobupivacaine for gynaecologic surgery

SECONDARY OUTCOMES:
side effects | 1 to 4 hours intraoperation plus within 2 hours in the recovery room
  to investigate side effects of intrathecal hyperbaric levobupivacaine compared with isobaric levobupivacaine for gynaecologic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vimolluck - Sanansilp, MD, Principal Investigator — Dept of Anesthesiology, Faculty of Medicine Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand